CLINICAL TRIAL: NCT02544464
Title: Does Intraoperative Intravenous Iron Enhance Postoperative Oxygenation Profile and the Recovery of Hemoglobin in Total Knee and Hip Arthroplasty Surgery?
Brief Title: Does Intraoperative Intravenous Iron Enhance Postoperative Oxygenation Profile in Total Knee Arthroplasty Surgery?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Collaborators: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KonkukUMC
Record Dates: First submitted 2015-09-03; First posted 2015-09-09 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; knee arthroplasty; iron
MeSH Terms: conditions — Osteoarthritis | interventions — ferric carboxymaltose; Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): ferric carboxymaltose 1000 mg
  Interventions: Drug: ferric carboxymaltose 1000 mg
- Control group (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ferric carboxymaltose 1000 mg — Ferric carboxymaltose is administered after anesthesia induction
  Other Names: Ferrinject
  Arms: Experimental group
Drug: placebo — placebo (normal saline) is administered after anesthesia induction
  Other Names: normal saline
  Arms: Control group

SUMMARY:
The objective of the present study is to determine the impact of intraoperative IV-iron supplementation on postoperative oxygenation profile by comparing the postoperative PaO2/FiO2 ratio with or without IV-iron supplementation in old patients undergoing elective uni-limb total knee arthroplasty surgery.

DETAILED DESCRIPTION:
Participation and recruitment: Patients undergoing elective total knee arthroplasty due to osteoarthritis will be interviewed for participation and recruited after providing written informed consent.

Randomization and group allocation:

All recruited patients will be given patient identification number (PIN) for the present study of 01-77 according to their order of interview and recruitment.

Investigators will prepare 33 yellow and 34 green cards, which will be inserted in 77 thick-paper envelopes. Then, all envelopes will be sealed, mixed and randomly allocated to get numbers of 01 to 77 (Envelop number).

After printing the envelope number outside envelope, all sealed envelopes with cards will be conveyed to and kept in pharmacy department.

Preparation and Administration of study drug:

Pharmacist will open the envelope with the number same to PIN and check the color of the card inside at study on operation day.

According to the color of the card, IV-iron or placebo will be prepared for the patient: IV-iron for yellow card; placebo for green cards, respectively.

The study drug was employed as "open labelled".

IV-iron or placebo will be infused through already established intravenous line within 30 min after anesthesia induction by attending anesthesiologist who is aware of the patient's group-allocation.

Patient data and statistical analyses:

The information regarding the patient's group allocation will be kept in the pharmacy department till the end of the study and conveyed during the data analyses after completion of the 77th patient participation and discharge.

Patient's data PaO2, FiO2, Hb, intra-op and postop-transfusion amount, intraop- and postop-bleeding amount will be determined from the patients' medical record after patient's discharge.

All statistical analyses will be performed after the 77th patient's discharge and data acquisition.

Surgical procedures:

All surgical procedures will be performed using standardized institutional anesthetic and surgical protocols, antibiotic and antithrombotic prophylaxis, transfusion protocols, and post-operative analgesia.

All TKA will be performed using a pneumatic tourniquet, which is deflated after wound closure. Closed suction drains, which are removed on the second post-operative day, will be placed in all operations.

Transfusion protocol:

Following allogenic blood transfusion protocol will be uniformly applied by anesthesiologists and surgeons to all patients in the operating theater, the post-operative anesthesia care unit, and the ward for the entire duration of hospitalization: blood transfusion of packed RBC will not be performed unless patient's Hb level is < 9 g/dL without any signs and/or symptoms of acute anemia such as hypotension, tachycardia, tachypnea, dizziness, and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis in knee joint undergoing elective uni-limb total knee arthroplasty surgery
* Patients provided a written informed consent.
* Patients with s-ferritin < 300 mg/dl (male) or 200 mg/dl (female)
* Patients with preoperative serum hemoglobin concentration >10 g/dL
* Patients with PaO2/FiO2 ratio >150

Exclusion Criteria:

* Patients with history of anaphylaxis, iron overload, active infection.
* Patients received or receiving intraoperative and preoperative blood salvaged, allogenic blood transfusion, recombinant human erythropoietin, or undergoing acute normovolemic hemodilution.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
The changes of Hemoglobin between preoperative and postoperative day 30 | postoperative 30 days
  intergroup-difference in hemoglobin change
the changes of arterial oxygen tension/inspired oxygen (PaO2/FiO2 ratio) | postoperative 5 days
  intergroup-difference in PaO2/FiO2 ratio

SECONDARY OUTCOMES:
arterial oxygen tension/inspired oxygen (PaO2/FiO2 ratio) | postoperative 1 day
  intergroup-difference in PaO2/FiO2 ratio
arterial oxygen tension/inspired oxygen (PaO2/FiO2 ratio) | postoperative 3 days
  intergroup-difference in PaO2/FiO2 ratio
arterial oxygen tension/inspired oxygen (PaO2/FiO2 ratio) | postoperative 5 days
  intergroup-difference in PaO2/FiO2 ratio
serum hemoglobin concentration | postoperative 1 day
  Intergroup difference of serum hemoglobin concentration, g/dL
serum hemoglobin concentration | postoperative 5 days
  Intergroup difference of serum hemoglobin concentration, g/dL
serum hemoglobin concentration | postoperative 30 days
  Intergroup difference of serum hemoglobin concentration, g/dL

CONTACTS AND LOCATIONS:
Locations (1):
- Konkuk University Medical Center & Asan Medical Center, Seoul, South Korea